CLINICAL TRIAL: NCT06853145
Title: Hyperpolarized Xenon-129 MRI in Idiopathic Pulmonary Fibrosis
Acronym: XeMRIIPF
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, John Kim, MD, MS, Medical Doctor, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HSR240022
Record Dates: First submitted 2024-11-01; First posted 2025-02-28 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-04

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Hyperpolarized Xenon-129 gas with MRI
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Intervention Model Description: IPF subjects will be scan via MRI using Hyperpolarized Xenon-129 gas
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- IPF subjects (Other): IPF subjects will undergo Xe-129 MRI
  Interventions: Drug: Hyperpolarized Xe129

INTERVENTIONS:
Drug: Hyperpolarized Xe129 — Hyperpolarized Xe129-MRI: Patients will undergo hyperpolarized Xe129-MRI at the University of Virginia Radiology Imaging Core (Charlottesville, VA, USA). The entire procedure visit takes approximately 3 hours based on our team's experience.
  Other Names: 129 HXe MRI

SUMMARY:
Idiopathic pulmonary fibrosis has a poor prognosis with limited treatment options. The Investigator hypothesize hyperpolarized Xe129-MRI can be performed in patients with IPF and repeated over time which will detect deficiencies related to perfusion in the lung.

DETAILED DESCRIPTION:
Idiopathic pulmonary fibrosis has a poor prognosis with limited treatment options. Idiopathic pulmonary fibrosis (IPF) is a subtype of interstitial lung disease (ILD) that can lead to chronic hypoxic and ventilatory respiratory failure and early death.1 While current treatments slow disease progression, they do not improve symptoms or quality of life and are often poorly tolerated due to significant side effect profiles. Therefore, there remains an unmet need for more tolerable therapies with an acceptable side effect profile that slows progression and improves patient-centered outcomes.

Functional imaging is a promising tool for assessing treatment response in IPF. Longitudinal decline in forced vital capacity (FVC) and time-to-event outcomes like hospitalization and death have been traditional clinical trial endpoints in IPF. However, these endpoints are time and resource-consuming. Thus, there has been significant interest in using other trial endpoints, the most promising of which is lung imaging. The study group employed hyperpolarized xenon-129 magnetic resonance imaging (Xe129-MRI) to quantify and localize deficits in pulmonary ventilation and perfusion in chronic obstructive diseases. It has recently extended this to pulmonary fibrosis. However, to implement Xe129-MRI as an endpoint in a mechanistic clinical trial, the investigator proposes to demonstrate the feasibility of employing this procedure over time in patients with IPF. The investigator hypothesizes that hyperpolarized Xe129-MRI can be performed in patients with IPF and repeated over time, which will detect deficiencies related to perfusion in the lung.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent 18 years of age or greater Clinical diagnosis of IPF

Exclusion Criteria:

* Continuous oxygen use at home
* Oxygen saturation less than 92% on the day of MRI procedure
* Pregnancy or lactation
* Claustrophobia, inner ear implants, aneurysm or other surgical clips, metal foreign bodies in eye, pacemaker or other contraindication to MR scanning. Subjects with any implanted device that cannot be verified as MRI compliant will be excluded.
* History of congenital cardiac disease, chronic renal failure, or cirrhosis. • Chest circumference greater than that of the xenon MR and/or helium coil. The circumference of the coil is approximately 42 inches.
* Inability to understand simple instructions or to hold still for approximately 10-15 seconds.
* History of respiratory infection within 2 weeks prior to the MR scan
* History of MI, stroke and/or poorly controlled hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Measuring the ventilation effect of HXe129 MRI for IPF subjects | Up to 24 hours post MR Imaging
  We will initially use descriptive statistics to describe the hyperpolarized Xe129 MRI indices and visualize their distribution using histograms. Paired t-test will be used to examine differences between baseline and follow-up hyperpolarized Xe129 MRI indices. Given that SA2 is to prove feasibility of accomplishing the MRI procedure, we have purposely opted to not adjust for the multiple MRI measurements that will be obtained.

SECONDARY OUTCOMES:
Measuring the diffusion capacity of HXe 129 for IPF subjects | Up to 24 hours post MRI analysis
  We will use linear mixed-effects model with random intercept and slope to determine the change in MRI indices over time between baseline and follow-up scans.

CONTACTS AND LOCATIONS:
Overall Officials: John Kim, MD, Principal Investigator — University of Virginia
Locations (1):
- Snyder Building 480 Ray C. Hunt Drive, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No